CLINICAL TRIAL: NCT06044870
Title: Clinical Evaluation of the Modified Laterally Stretched Technique in the Gingival Recession Sites of the Lower Anterior Teeth (RT2) vs Tunneling With Connective Tissue Grafting in Both Techniques: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of the Modified Laterally Stretched Technique (RT2) Gingival Recession vs Tunneling With CT Grafting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha fawzy el sayed ali abd allah, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21021992
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified laterally stretched technique with a connective tissue graft. (Experimental): After the administration of local anesthesia, root planing of the exposed root surfaces will be performed by means of hand instruments.
  A partial thickness envelope is performed with tunneling instruments involving one or two teeth adjacent to the tooth, in case of a very thin biotype a complete thickness envelope could be done.
  Two horizontal incisions are done at the base of the papillae of the deepest recession site, allowing to place the graft in a more coronal position and improving access and visibility.
  Interventions: Procedure: Modified laterally stretched technique with a connective tissue graft.
- Tunneling technique with connective tissue graft. (Active Comparator): Immediately before surgery, contact point composite stops were placed to prevent the collapse of the suspended sutures in the inter-proximal spaces.• The entire gingival papillary complex will be moved coronally using a suspended suture anchored in the lingual gingiva (Aroca et al., 2010, 2013; Azzi et al, 2002, zuhr et al.,2009).
  Interventions: Procedure: Modified laterally stretched technique with a connective tissue graft.

INTERVENTIONS:
Procedure: Modified laterally stretched technique with a connective tissue graft. — Modified laterally stretched technique with a connective tissue graft.

SUMMARY:
Regression analysis in a recent systematic review showed significantly greater mRC and CRC values when modifications are done to the TUN procedure to achieve more coronal advancement of the flap, coronal advancement also helps in covering the underlying graft for better recession coverage outcomes (Tavelli et al., 2018), limited data is present on the possible influence of a covered or partially uncovered graft. However, it has been suggested that minimal exposure of the CTG may aid not only in achieving CRC but also a harmonious gingival margin (John et al., 2015; Rasperini et al., 2011).

ELIGIBILITY:
* Single or multiple RT2 gingival recession site/sites in the lower anterior teeth.
* Age >/= 18 years.
* Patients with healthy or treated periodontal conditions.
* Patients willing to participate in the study.
* Absence of uncontrolled medical conditions.
* Full mouth plaque score </= 20% (O'Leary 1972).
* Full mouth bleeding score <20% (Ainamo and Bay 1975).
* Patients with aesthetic concerns.

Exclusion Criteria:

* Pregnant or lactating females.
* deep recession sites more than 5 mm
* Tobacco smoking.
* Uncontrolled medical conditions.
* Uncooperative patients or unable to complete the study.
* Patients treated with any medication known to cause gingival hyperplasia.
* No occlusal interferences.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Recession depth reduction. | 1 year
  Measured as the difference between the recession gingival depth at different follow up intervals and the baseline.

SECONDARY OUTCOMES:
Mean root coverage | 1 year
  (Preoperative vertical recession - Postoperative vertical recession/preoperative vertical recession) x 100
Recession depth | 1 year
  Measured as the distance between the free gingival margin and the cemento-enamel junction .
Recession width | 1 year
  Measured as the distance between the between the mesial gingival margin and distal gingival margin
Soft tissue thickness | 1 year
  The measurement of Gingival tissue thickness is performed 2 mm apical from the gingival margin.
Keratinized tissue width | 1 year
  Measured as the distance between the gingival margin and the muco-gingival junction.
Esthetics (RES) score | 1 year
  A system used to evaluate five variables 6 months gingival margin (GM), marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC).
patient satisfaction | 1 year
  A 3-item questionnaire is asked, and the patients shall use a 7-point answer scale. The answers were given on a 7-point scale ranging from 1 'not at all'' to 7 ''very likely''.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No